CLINICAL TRIAL: NCT01883336
Title: Long Term Follow up of Small Non-inflammatory Pancreatic Cysts - a Retrospective Multicenter Study.
Brief Title: Long Term Follow up of Small Non-inflammatory Pancreatic Cysts
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Prof. Dr. Thomas Roesch, Universitätsklinikum Hamburg Eppendorf, Endoscopy department, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: UKE HH Endoscopy PV3879
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cysts
Keywords: Incidental pancreatic cysts
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study intends to investigate the long term follow-up of small non-inflammatory pancreatic cysts.

DETAILED DESCRIPTION:
This study intends to investigate the long term follow-up of small non-inflammatory pancreatic cysts in a multicenter setting.

Inclusion criteria:

Patients with non-inflammatory pancreatic cystic lesions up to 3 cm in diameter referred to the University Hospital Hamburg Eppendorf, Israelitic Hospital Hamburg, Sana Klinikum Lichtenberg, Berlin and Krankenhaus Märkisch-Oderland,Strausberg from 2002 to 2007 identified from EUS database.

Study design:

At least 5 year-long term follow up by inclusion of clinical data, cross sectional imaging if available or actual US findings.

Primary outcome:

To determine the proportion of patients with increase is size and/or changed appearance

Secondary outcomes:

Rate of patients undergo pancreatic surgery (indication, histology of resected specimen). Rate of patients undergo FNA (fluid analysis, cytology).

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-inflammatory pancreatic cystic lesions up to 3 cm in diameter

Exclusion Criteria:

* acute or chronic pancreatitis
* pancreatic cysts > 3 cm
* Lesion suspicious for malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-inflammatory pancreatic cystic lesions up to 3 cm in diameter referred to the University Hospital Hamburg Eppendorf, Israelitic Hospital Hamburg, Sana Klinikum Lichtenberg, Berlin and Krankenhaus Märkisch-Oderland,Strausberg.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Progress of pancreatic cyst | 5 years
  To determine the proportion of patients with increase is size and/or changed appearance of pancreatic cyst.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roesch, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany